CLINICAL TRIAL: NCT00115726
Title: Randomized Controlled Trial Assessing the Effect of Preoperative Furosemide on Intraoperative Blood Pressure
Brief Title: Trial Assessing the Effect of Preoperative Furosemide on Intraoperative Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Centre for the Advancement of Health (Unknown)
Responsible Party: Dr. Nadia Khan, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15326; 15326
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Hypertension; Hypotension; Edema; Congestive Heart Failure
Keywords: anesthesia; hypotension; furosemide; blood pressure; peripheral edema; diuretic; surgery; congestive heart failure
MeSH Terms: conditions — Hypertension; Hypotension; Edema; Heart Failure | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): furosemide
  Interventions: Drug: furosemide
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: furosemide — for patients on chronic furosemide therapy, patients are randomized to furosemide (at their previous dose) or placebo (given in identical form to ensure masking)
  Arms: 1
Drug: placebo — patients will be given placebo capsules (identical to experimental arm in color) at the equivalent dose as to their chronic furosemide therapy.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether continuing or discontinuing furosemide (a diuretic) on the day of elective noncardiac surgery for those who take furosemide on a chronic basis, causes more intraoperative hypotension (low blood pressure) during surgery. Our hypothesis is that the usual practice of continuing furosemide on the day of surgery would contribute to more hypotension during surgery than discontinuing furosemide.

DETAILED DESCRIPTION:
A significant proportion of patients who undergo surgery take medications on a chronic basis. Little is known about the effects of these medications on the successful conduct of anesthesia and surgery. Diuretics like furosemide may contribute to low blood pressure during surgery, an outcome associated with cardiovascular complications. However, many patients are recommended to take their diuretics on the day of surgery. We wished to determine if preoperative administration of furosemide contributes to intraoperative hypotension compared to placebo.

Comparison: We conducted a randomized, double blind placebo controlled trial to compare the effect of furosemide with that of placebo on intraoperative hypotension using intraoperative blood pressure recordings in patients who take furosemide chronically and were undergoing noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adults referred to preoperative assessment clinics by surgeons for elective non-cardiac surgery who routinely take furosemide.
* Participants must also be able to give informed consent

Exclusion Criteria:

* Less than 18 years of age
* Have comorbid conditions with which brief periods of hypotension may be particularly harmful such as: 1) pregnancy; 2) baseline hypotension (systolic <100 mmHg at the preoperative assessment clinic); 3) autonomic dysfunction; 4) severe aortic stenosis.
* Patients who take furosemide only on an 'as needed basis' rather than 'regularly'.
* Those patients who take less than 10 mg of furosemide daily
* Those patients who are undergoing local anesthetic only surgical procedures
* Patients who are unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2000-09; Primary Completion 2006-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing hypotension during the operative period. Hypotension is defined based on blood pressure criteria (systolic BP <90 mmHg or 35% drop in mean arterial pressure) (or vasopressor treatment during surgery). | hospital stay

SECONDARY OUTCOMES:
Patients will be followed up for the duration of their hospital stay for the following endpoints: (1) Development of congestive heart failure exacerbation | hospital stay
(2) Total cardiovascular complications: composite of acute myocardial infarction, angina, stroke/TIA, arrhythmia, congestive heart failure or cardiac death. | hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Norman RC Campbell, MD, Principal Investigator — University of Calgary, Calgary, Alberta, Canada
Locations (3):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States
- Canada (2):
  - Foothills Hospital, Calgary, Alberta
  - University of Western Ontario, London, Ontario